CLINICAL TRIAL: NCT01637038
Title: The Effect of Remote Ischemic Postconditioning on Liver Graft and Renal Function in Patients Undergoing Living-related Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2012-06-010-001
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Ischemia/Reperfusion Injury of Liver Graft; Ischemia/Reperfusion Injury of Kidney; Remote Ischemic Postconditioning
Keywords: ischemia/reperfusion injury; remote ischemic postconditioning
MeSH Terms: conditions — Ischemia; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): no intervention
- RIPC group (Experimental): Those undergoing remote ischemic postconditioning
  Interventions: Other: RIPC

INTERVENTIONS:
Other: RIPC — Those undergoing remote ischemic postconditioning. Remote ischemic postconditioning consists of three 5-min cycles of upper limb ischemia, which was induced by an automated cuff-inflator placed on the unilateral upper limb and inflated to 250 mm Hg, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Other Names: remote ischemic postconditioning
  Arms: RIPC group

SUMMARY:
The investigators are trying to evaluate the clinical effect of remote ischemic postconditioning on liver graft function and postoperative renal function in subjects undergoing living-donor liver transplantation.

DETAILED DESCRIPTION:
Ischemic reperfusion injury of liver graft and postoperative renal dysfunction is a common problem which influence poor outcome in subjects undergoing liver transplantation. The incidence of postoperative renal dysfunction was reported as high as 12 ~ 64% and is thought to be caused by ischemia/reperfusion injury. Ischemic pre- or postconditioning was reported to be effective for preventing ischemia/reperfusion injury during liver transplantation. Remote ischemic pre- or postconditioning was also reported to be protective for ischemia/reperfusion injury in major organs in previous animal studies. Therefore, we are trying to evaluate the clinical effect of remote ischemic postconditioning on liver graft function and postoperative renal function in subjects undergoing living-donor liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing living donor liver transplantation during the study period
* Subjects older than 20 yrs who can give written informed consent

Exclusion Criteria:

* Re-transplanted recipients
* Those with peripheral vascular diseases affecting the extremities
* Those with hepatic encephalopathy
* Those with cirrhotic cardiomyopathy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
total bilirubin | before surgery and at 6, 12, 24, 36, 48, 60, 72, 84, 96 hours after the end of surgery
  total bilirubin before surgery and at 6, 12, 24, 36, 48, 60, 72, 84, 96 hours after the end of surgery

SECONDARY OUTCOMES:
Renal Function Test profiles | Before surgery and at 6, 12, 24, 36, 48, 60, 72, 84, 96 hours after the end of surgery
  Serum BUN, creatinine concentration, estimated GFR and urine output before surgery and at 6, 12, 24, 36, 48, 60, 72, 84, 96 hours after the end of surgery
Liver Function Test Profiles | before surgery and at 6, 12, 24, 36, 48, 60, 72, 84, 96 hours after the end of surgery
  AST, ALT, albumin, before surgery and at 6, 12, 24, 36, 48, 60, 72, 84, 96 hours after the end of surgery
incidence of Surgical Outcome | 1 week, 1 month after the end of surgery
  incidence of acute rejection of transplanted Liver (Biopsy-confirmed or clinically symptomatic),incidence of Delayed graft function : clinically symptomatic, incidecne of Postoperative renal replacement therapy
Length of hospital stay (days) | 1 month, 2 month, 3 month after the end of surgery
  total hospital stay, ICU stay, postoperative stay

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hwan Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea